CLINICAL TRIAL: NCT01455987
Title: Outcome of the Knee Osteochonditis Dissecans Patiets in Kuopio University Hospital (1990-2009): A Retropective Analysis
Brief Title: Osteochondritis Dissecans of the Knee
Acronym: KYSOCD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Pekko Penttila, M.D. Postgraduate student. Resident in Pediatric Surgery, Kuopio University Hospital
Other Study IDs: KUH5203050
Record Dates: First submitted 2011-01-04; First posted 2011-10-20 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Osteochondritis Dissecans; Juvenile Osteochondritis Dissecans
Keywords: Osteochondritis dissecans; Juvenile osteochondritis dissecans; Knee; Osteochondral; Outcome
MeSH Terms: conditions — Osteochondritis Dissecans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Osteochondritis dissecans is a relatively common...

ELIGIBILITY:
Inclusion Criteria:

* Osteochondritis dissecans diagnosis code (ICD-8 to -10) in the medical records of KUH
* Knee OCD verified from the medical records

Exclusion Criteria:

-Any other medical condition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been treated in Kuopio University Hospital (KUH) district for osteochondritis dissecans of the knee between 1.1.1990 and 31.12.2009.
Sampling Method: Probability Sample
Enrollment: 265 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Knee pain measured by NRS (numeric rating scale, 0-10) | At the time of recruiting, which is an avarage calculated from all participiants enrolled for this study (estimated avarage follow-up 12-16 years).
  0=no pain 10=maximal pain

SECONDARY OUTCOMES:
Lysholm Knee Score and Knee Injury and Osteoarthritis Outcome Score (KOOS) | At the time of recruiting, which is an avarage calculated from all participiants enrolled for this study (estimated avarage follow-up 12-16 years).
  Lysholm Knee Score and KOOS are validated subjective questionares assessing outcome after knee surgery/injury.